CLINICAL TRIAL: NCT04135768
Title: A Prospective, Randomised Controlled Pilot Trial Of Wrist Joint Haematoma Washout As An Adjunct To Volar Plating In Intra-articular Distal Radius Fractures
Brief Title: A Study Examining The Effect Of Wrist Joint Haematoma Washout As An Adjunct Procedure To Plating Of The Distal Radius In Fractures Of The Distal Radius Involving The Wrist Joint
Acronym: JWDRF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 pandemic: national lockdown imposed and study centre diverted all trauma cases to surrounding hospitals
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Ong Jo Hann, Orthopaedic Trainee, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Radius Fracture Distal
Keywords: Distal radius fracture; Articular fracture; Joint haematoma; Volar wrist plating
MeSH Terms: conditions — Wrist Fractures; Intra-Articular Fractures

STUDY DESIGN:
Intervention Model Description: Pilot study, single center, parallel group design
Who Masked: Participant
Masking Description: Participants are blinded, since the study procedure will be performed via the incision for the main surgery. Thus no external (wound) evidence of the participant's allocation will be visible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants who will undergo both volar locking plate fixation of the distal radius and the study procedure (wrist joint haematoma washout)
  Interventions: Procedure: Wrist joint haematoma washout; Procedure: Volar locking plate insertion of the distal radius
- Placebo (Placebo Comparator): Participants who will undergo volar locking plate fixation of the distal radius only
  Interventions: Procedure: Volar locking plate insertion of the distal radius

INTERVENTIONS:
Procedure: Wrist joint haematoma washout — After plating of the distal radius is performed, a small incision is made on the wrist joint capsule. This is the portal for fluid efflux. An intravenous cannula is used to puncture the wrist joint capsule adjacent to the first incision and normal saline is infused through this cannula into the wrist joint. The infusion continues until the fluid efflux from the first portal is clear and no longer blood stained. This will be the point at which the washout is considered to be complete.
  Arms: Treatment
Procedure: Volar locking plate insertion of the distal radius — An anatomical locking plate is applied to the distal radius fracture using screws

SUMMARY:
Intra-articular fractures of the distal radius are common in urban populations and result in significant morbidity in terms of time away from work. Volar plating of the distal radius is a commonly used mode of surgical fixation of this fracture. The joint haematoma resulting from the fracture has been hypothesized to contribute to the post-injury disability. As such, this study aims to examine if the evacuation of the haematoma during volar plating results in superior functional outcomes at three months post surgery.

DETAILED DESCRIPTION:
Distal radius fractures have an incidence of up to 50% of all fractures, with up to two thirds being intra-articular fractures. While most fractures treated with a variety of methods achieve satisfactory patient reported outcomes at one year post treatment, patients experience pain and functional impairment up to 3 and 6 months post treatment. Open reduction and internal fixation using volar plates is one popular mode of treatment. It is relatively widely available and allows almost immediate post operative mobilisation and rehabilitation.

One theory which could explain the delay in functional recovery is the persistence of the intra-articular haematoma. The evacuation of this haematoma may be partly responsible for the satisfactory results published by authors who perform wrist arthroscopy assisted distal radius fixation.

In our literature review, it is not routine to evacuate this haematoma during conventional volar plating of the distal radius. As such, we aim to study if the evacuation of the haematoma in conjunction with volar plating confers functional benefits in the short term, particularly at 3 months post surgery.

ELIGIBILITY:
INCLUSION CRITERIA:

Skeletally mature patients of either sex who sustain closed fractures of the distal end radius involving the articular surface, between the ages of 18 and 65

The fracture pattern is of an unacceptable morphology as defined by the following radiographic parameters according to the 2009 American Academy of Orthopaedic Surgeons (AAOS) Clinical Guidelines (Lichtmann, Bindra et al. 2010):

>3 mm radial shortening >10° dorsal tilt >2 mm articular displacement The patient has been planned to undergo VLPF Femalepatientswilleitherbe Post-menopausal Surgically sterile If of childbearing age, must have a negative urine pregnancy test at screening and at randomisation. Pregnancy tests will be repeated during each visit.

EXCLUSION CRITERIA:

Open fractures Associated fractures around the wrist (e.g. carpal bones, metacarpals, phalanges) requiring different or additional methods of fracture fixation and stabilisation Polytraumatised patients Compartmentsyndromeoftheforearmorhand Neurovascular injury of the ipsilateral limb Concomitantfractureoftheipsilateraland/orcontralateralupperlimbwhichmayimpede post-operative rehabilitation Fractures exceeding 14 days duration during time of first presentation

Pre-existing conditions such as:

Inflammatory arthritides Connective tissue diseases Diseases of bone metabolism (except osteoporosis) Prior malunited/nonunited fractures of the ipsilateral limb Pregnancy Patients unfit for surgery due to poor general condition Inability or unwillingness to provide written consent. Inability or unwillingness to comply with the requirements of the protocol as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference between QuickDASH scores of both treatment arms at 3 months | 3 months
  A patient reported outcome using the QuickDASH (Quick Disabilities of the Arm, Shoulder and Hand) score. This is a patient reported outcome score, which consists of 11 questions. A minimum of 10 must be answered for the score to be valid. The score out of 11 is then calculated as a percentage, with higher numbers indicating worse disability.

SECONDARY OUTCOMES:
Mean difference between QuickDASH scores of both treatment arms at 2 weeks, 6 weeks, and 6 months | 2 weeks, 6 weeks and 6 months
  Comparing patient reported outcomes at other points of time in follow up. This is a patient reported outcome score, which consists of 11 questions. A minimum of 10 must be answered for the score to be valid. The score out of 11 is then calculated as a percentage, with higher numbers indicating worse disability.
Mean difference of rate of improvement of QuickDASH scores between groups across 6 months of follow up | 6 months
  Assessing difference in rate of change of the QuickDASH score over time.This is a patient reported outcome score, which consists of 11 questions. A minimum of 10 must be answered for the score to be valid. The score out of 11 is then calculated as a percentage, with higher numbers indicating worse disability.
Mean difference between the visual analogue scores of both groups | 2 weeks, 6 weeks, 3 months and 6 months
  Visual analogue scores of pain (out of 10). Higher scores indicate more severe pain.
Mean difference between the grip strength of both groups | 2 weeks, 6 weeks, 3 months and 6 months
  Grip strength as measured by a Jamar dynamometer, described as a percentage of the uninjured limb
Mean difference between the range of motion of the wrist of both groups | 2 weeks, 6 weeks, 3 months and 6 months
  Assessing range of motion in flexion, extension, pronation, supination, radial deviation and ulnar deviation
Mean difference between rate of complications of both groups | 6 months
  Complications such as infection, tendon irritation/rupture/adhesions, complex regional pain syndrome, etc
Mean difference in time to radiographic fracture union of both groups | 6 months
  Assessing X rays at follow up to determine radiographically that the fracture is united. This is determined as the point at which at least 3 out of 4 cortices of the fracture are bridged with callus on two orthogonal X ray views of the wrist

CONTACTS AND LOCATIONS:
Overall Officials: Tunku Sara Tunku Ahmad Yahaya, FRCS, Study Chair — University of Malaya Medical Center
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Participant results only will be made available to other researchers from University of Malaya should a related study be conducted. Identifying data will not be shared. Participants will be identified by subject ID only

REFERENCES:
- [Background] Abe Y, Fujii K. Arthroscopic-Assisted Reduction of Intra-articular Distal Radius Fracture. Hand Clin. 2017 Nov;33(4):659-668. doi: 10.1016/j.hcl.2017.07.011. PMID 28991578
- [Background] MacDermid JC, Roth JH, Richards RS. Pain and disability reported in the year following a distal radius fracture: a cohort study. BMC Musculoskelet Disord. 2003 Oct 31;4:24. doi: 10.1186/1471-2474-4-24. PMID 14588078
- [Background] Smeraglia F, Del Buono A, Maffulli N. Wrist arthroscopy in the management of articular distal radius fractures. Br Med Bull. 2016 Sep;119(1):157-65. doi: 10.1093/bmb/ldw032. Epub 2016 Aug 22. PMID 27554281
- [Background] Gouk CJC, Bindra RR, Tarrant DJ, Thomas MJE. Volar locking plate fixation versus external fixation of distal radius fractures: a meta-analysis. J Hand Surg Eur Vol. 2018 Nov;43(9):954-960. doi: 10.1177/1753193417743936. Epub 2017 Dec 11. PMID 29228851